CLINICAL TRIAL: NCT06583785
Title: Impact of Anthocyanin-Rich Black Rice Consumption on Cognitive Function, Inflammation and Micro-vascular Function in Older Adults
Brief Title: Black Rice Consumption on Cognitive Function, Inflammation and Microvascular Function in Older Adults
Acronym: RICE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Jeremy Paul Edward Spencer, Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: UREC 23/30
Record Dates: First submitted 2024-05-15; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Older Adults
Keywords: Cognitive function; Inflammation; Memory; Older adults
MeSH Terms: conditions — Inflammation | interventions — Methods

STUDY DESIGN:
Intervention Model Description: A randomized, open-label, crossover design with a week wash-out period for investigating the acute and short-term effects of black rice consumption on the cognitive function, inflammation and microvascular function in older adults.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Black rice (Experimental): Black rice (210g/meal). Acute study: the volunteers will be asked to eat black rice meal and measured outcomes at 2 hours after consumption.
  Short-term study: the volunteers will be asked to consume black rice meals for 7 consecutive days.
  Interventions: Other: Black rice (Intervention); Other: Brown rice (Control)
- Brown rice (Placebo Comparator): Brown rice (210g/meal). Acute study: the volunteers will be asked to eat brown rice meal and measured outcomes at 2 hours after consumption.
  Short-term study: the volunteers will be asked to consume brown rice meals for 7 consecutive days.
  Interventions: Other: Black rice (Intervention); Other: Brown rice (Control)

INTERVENTIONS:
Other: Black rice (Intervention) — 210 g of cooked black rice
Other: Brown rice (Control) — 210 g of cooked brown rice

SUMMARY:
Cognitive (brain) function, especially memory, gradually declines during ageing, which may in part be caused by an increase in systemic inflammation as well as a reduction in vascular functions and cerebral blood flow. Blood inflammatory mediators such as c-reactive protein (CRP) and interleukin-6 (IL-6) found to be significantly higher among people over 65 years compared to younger age groups.

Anthocyanins is water-soluble compounds giving blue, purple and red colours in fruits and vegetables. Anthocyanins have been demonstrated to improve cognitive function, inhibit inflammation, and protect cardiovascular health. Black rice contains high amounts of anthocyanins mainly cyanidin 3-glucoside and peonidin 3-glucoside as well as various nutritional compounds such as carbohydrate, vitamin B, vitamin E and fibre. Previous studies reported health benefits of black rice, including anti-inflammation, antioxidative stress, anti-diabetes, and improved cognitive function. However, the effect of black rice consumption on cognitive function related to inflammation has not been studied in humans.

Therefore, this study aims evaluate the acute & short-term effects of black rice consumption on the cognitive function, inflammation, and vascular function in older adults aged 50-80 years.

The primary and secondary research questions of this study will address:

1. Do the acute and short-term anthocyanin-rich black rice intakes improve cognitive function in older adults aged 50-80 years?
2. Do the acute and short-term anthocyanin-rich black rice intakes modulate inflammatory status and microvascular function in older adults aged 50-80 years?

DETAILED DESCRIPTION:
This study is a randomised controlled crossover design with a week wash-out period for investigating the acute (2 hrs), short-term (7 days), and acute on short-term (7 days, 2 hrs) effects of black rice consumption on the cognitiv function, inflammation, and vascular function in older adults aged 50-80 years. The cognitive function will be assessed using computer-based test via Gorilla platform. The inflammatory mediators will be measured in a blood sample. The vascular function will be tested by Laser Doppler imaging with iontophoresis (LDI), blood pressure (BP) and heart rate (HR).

Eligible volunteers will be asked to attend the Hugh Sinclair Unit of Human Nutrition for 1 screening visit and 4 study visits.

The enrolment, volunteers will be recruited by poster, E-mail, or telephone. If they are interested in the study and meet the criteria, volunteers will be provided with the participant information sheet explaining the nature and requirements of study. The volunteers who are interested in attending the study will be asked to fill out the health and lifestyle screening questionnaires online link. The potentially eligible volunteers will be invited to attend a screening visit at the Hugh Sinclair Unit of Human Nutrition.

For screening visit (approximately 1-1.5 h), the researcher will explain all the details of the study to volunteers and confirm information in a screening questionnaire. The volunteers who meet the study criteria will be asked to sign the informed consent before partaking in the study. Height, weight, waist circumference, BP, and HR will be measured. Then, global cognitive performance (MMSE test) will be assessed. Inclusion/exclusion criteria will then be reviewed for participant eligibility. Then, they will be asked to perform the demo cognitive tests (30 min). The volunteers will be provided with the participant information booklet which contains the guidelines on what to do during the study and will be invited to attend the study in following week. the volunteers will be asked to fill out food frequency questionnaire prior to first visit.

For study visit 1-4, the volunteers will be asked to fast 8 hours in advance. They will be asked to consume a low the polyphenol rich diet for 24 hours in advance of 1st and 3rd study visit. As soon as they arrive at the nutritional unit, the 15 ml of venous blood will be taken, followed by cognitive testing and BP, HR and LDI will be completed at baseline (35-40 min). After that, the volunteers will receive cooked black rice or control cooked brown rice in a random order served with omelette and 1 glass of water. The volunteers will be asked to eat tested meal within 20 minutes. Then, 2 hours after consumption, the cognitive function will be then assessed, followed by LDI, BP and HR measurements.

For the short-term intervention (to be continued after 1st and 3rd study visit), the volunteers will be provided raw rice and a rice cooker for cooking at home for a further 7 days. The volunteers will be asked to have daily rice consumption (1 meal per day) with avoiding anthocyanin rich food but maintain habitual physical activity during study. In addition, they will be asked to do daily check list to confirm study compliance during trial.

A power calculation based on three similar studies investigating the acute effect of anthocyanin-rich food consumption on cognitive function in middle aged-older adults which suggested that 24 participants (include 10% attribution rate) should provide the sufficient statistic power (Average Effect size=0.64, α=0.05, Power=0.8).

the collected data will be anonymised by providing each participant with unique identification number. The key file will be stored securely in a password protection folder stored in the University-managed cloud. Following completion of the study, the data will be fully anonymised before being archived. Only the applicants named on this form will be digital access to the data and only the researchers directly related to the study will have physical access to keys to the filing cabinets where the paper forms will be stored.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50-80 years
* General healthy status
* Body Mass Index (BMI)18.5-35 kg/m2

Exclusion Criteria:

* Taking anti-inflammatory drugs (e.g., aspirin, warfarin, ibuprofen)
* Having sign of infections or acute inflammation (e.g., fever, chills, sore throat, nasal congestion, moderate-severe pain, swelling-redness)
* Received antibiotics within the past 3 months
* Taking dietary supplements (e.g., vitamins, minerals) at high doses (e.g., more than 200% of the UK's reference nutrient intakes)
* Taking hormone replacement therapy, if you are menopausal
* Had major surgery (head, heart, chest, abdomen) within the past 6 months.
* Having plan to start to a restricted diet/ changing dietary pattern or lose weight.
* Diagnosed with neurodegenerative diseases (e.g., Dementia, Alzheimer's, Parkinson's, current stroke)
* Diagnosed with psychotic disorders (e.g., schizophrenia, bipolar depression, eating disorder)
* Diagnosed with cardiovascular disease, diabetes, hyperlipidemia, hypertension (blood pressure>140/90 mmHg), active cancer, liver, or kidney diseases.
* Taking medication to lower blood fats (e.g., statins, fibrates) or to stabilise blood glucose (e.g., acarbose, metformin or sulfonylureas) or lower blood pressure.
* Unable to complete the cognitive function tasks for any reason (i.e., visual impairments, hearing loss)
* If you have a peacemaker
* If you have bleeding disorders or blood related diseases (anaemia, thalassemia, thrombosis, embolism)
* Heavy smoker
* Heavy alcohol drinking (> 14 units/week) or a history of alcohol/substance abuse
* Allergies, hypersensitivity, or food intolerances (rice, eggs, soy sauce, vegetable oil)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rey Auditory Verbal Learning (RAVLT) | Day 0, 2hrs, Day 7, Day 7-2hrs
  This task consists of 5 consecutive free recalls of the same 15 nouns presented as a first auditory list (list A), followed by recall of a further 15 nouns presented as an interference list (list B) which is recalled only once. After 15 words had been presented, participants will be asked to say aloud each word as many as they can recall in any order (approximately a minute). The session will be occurred five times. Then, the participants listen an auditory list of 15 words (list B) and will be asked to say aloud each word as many as they can recall in any order. The number of correct words will be counted and averaged of five trials (list A).
  Measurements: at baseline (Day 0), acute intervention (2hrs), 7 days short-term intervention (Day 7) and acute on short-term intervention (Day7-2hrs)
Digit span Forward and Backward tasks | Day 0, 2hrs, Day 7, Day 7-2hrs
  In this task, the series of digits (numbers) of varying length (spans of 2-9 for forward and 2-8 for backward). It consists of 8 items of forward and 7 items of backward tasks and has 2 trials for each item. The forward and backward digit span tasks, the number will be presented on computer screen an increasingly longer series of digits at a rate of 1 digit/s. The participants will be asked to repeat the number by pressing number on the keyboard. The score will be the maximum of digits of correct both trials, prior to failing two consecutive trials at any one span size.
  Measurements: at baseline (Day 0), acute intervention (2hrs), 7 days short-term intervention (Day 7) and acute on short-term intervention (Day7-2hrs)
Stroop task | Day 0, 2hrs, Day 7, Day 7-2hrs
  The participants were presented with the words 'GREEN', 'BLUE', 'RED' and 'YELLOW', which were displayed either in the same colour ink as the meaning of the word (congruent trials) or in a colour inconsistent with the meaning of the word (incongruent trials). The participant will be instructed to respond to the colour in which the word is presented rather than the meaning of the word, by pressing a corresponding key on the keyboard. There were 96 trials in total and the task lasted for approximately four minutes. The primary dependent variable was reaction time for correct responses.
  Measurements: at baseline (Day 0), acute intervention (2hrs), 7 days short-term intervention (Day 7) and acute on short-term intervention (Day7-2hrs)
The Digit Symbol-Substitution Task (DSST) | Day 0, 2hrs, Day 7, Day 7-2hrs
  Participants are given a table pairing the digits 1 through 9 with nine distinct symbols. Below the table, there is four rows of 25 boxes, each containing a number from one to nine with a blank box underneath. The numbered boxes will be in a random order. Starting at the beginning of the first row and working from left to right down the page, participants will be asked to fill the correct symbol in the blank box using the key at the top of the page. Participants were given 90 seconds to fill in as many boxes as possible in sequential order and the total number of correctly completed boxes will be used to indicate processing speed.
  Measurements: at baseline (Day 0), acute intervention (2hrs), 7 days short-term intervention (Day 7) and acute on short-term intervention (Day7-2hrs)

SECONDARY OUTCOMES:
High sensitive C reactive protein (hs-CRP) | Day 0, Day 7
  Serum hs-CRP (mg/L) will be analyzed by automated Enzyme immunoassays (ELISA).
Serum inflammatory markers | Day 0, Day 7
  All serum inflammatory markers including, IL-6 (pg/ml), IL-1β (pg/ml), and TNF-α (pg/ml) will be analyzed by automated Enzyme immunoassays (ELISA).
Laser Doppler imaging (LDI) | Day 0, 2hrs, Day 7, Day 7-2hrs
  The microvascular blood flow will be measured by LDI technique which assesses the changing of skin blood flow in response to acetylcholine and sodium nitroprusside by iontophoresis.
Blood pressure (BP) | Day 0, 2hrs, Day 7, Day 7-2hrs
  BP (mmHg) will be measeured by Omron BP monitor.
Heart rate (HR) | Day 0, 2hrs, Day 7, Day 7-2hrs
  HP (beat per minute, BPM) will be measeured by Omron BP monitor.
Vascular cell adhesion protein 1 (VCAM-1) | Day 0, Day 7
  Serum VCAM-1(ng/ml) will be analyzed by automated ELISA.
Intercellular adhesion molecule-1 (ICAM-1) | Day 0, Day 7
  Serum ICAM-1 (ng/ml) will be analyzed by automated ELISA.
Brain-derived neurotrophic factor (BDNF) | Day 0, Day 7
  Serum BDNF (pg/ml) will be analyzed by automated ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Spencer, PhD, Principal Investigator — Department of Food and Nutritional Sciences, University of Reading
Locations (2):
- United Kingdom (2):
  - Hugh Sinclair Unit of Human Nutrition, Reading, UK
  - Hugh Sinclair Unit of Human Nutrition, Department of Food and Nutritional Sciences, University of Reading, Reading

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mekhora C, Lamport DJ, Spencer JPE. Impact of anthocyanin-rich black rice consumption on cognitive function, inflammation and microvascular function in older adults: a crossover intervention trial. Food Funct. 2026 Jan 13. doi: 10.1039/d5fo04351d. Online ahead of print. PMID 41528201